CLINICAL TRIAL: NCT05582070
Title: Effect on Sleep of Surgical Treatment of Severe Nasal Obstruction
Acronym: SOMNOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2022/15
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Sleep Apnea; Obstructive Sleep Apnea; Nasal Obstruction
Keywords: OSA; sleep apnea; nasal surgery; nasal desobstruction; sleep quality; actigraphy; wake after sleep onset; WASO
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Nasal Obstruction; Sleep Initiation and Maintenance Disorders | interventions — Actigraphy

STUDY DESIGN:
Intervention Model Description: prospective, monocentric study, non-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- actigraphy (Experimental): Patient with nasal obstruction
  Interventions: Other: actigraphy

INTERVENTIONS:
Other: actigraphy — Actigraphy examination will be performed during 2 periods of 7 days before and after nose nasal desobstruction surgery (septoplasty, septorhinoplasty or total ethmoidectomy). Respectively 2 months before surgery (inclusion) and 4 months after surgery.

SUMMARY:
The aim of the study is to evaluate the effect of nasal desobstruction surgery (septoplasty, septorhinoplasty or total ethmoidectomy) on sleep quality, assessed by the variation of the Wake after sleep onset (WASO), in patients presenting with sleep disorders and severe nasal obstruction.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSA) is a sleep breathing disorder characterised by episodes of complete or partial obstruction of the upper airway. OSA is a common disease which impacts quality of life, mood, cardiovascular morbidity, and mortality. It is often under-diagnosed and is estimated to affect at least 2-5% of the female population and 3-7% of the male population.

Currently, nasal obstruction is not recognised as an independent risk factor for obstructive sleep apnea syndrome. The current definition of OSA is based on an Apnea/Hypopnea index (AHI) greater than five. However, most studies do not find a decrease in this index after nasal desobstruction surgery despite a significant improvement in sleep quality scales. The AHI index appears to be a limited paraclinical criteria to assess the impact of nasal obstruction on sleep quality.

Other objective paraclinical criteria have been used in other nosological sleep settings to objectively assess sleep quality. These include the WASO (wake after sleep onset) criteria. To investigators knowledge, no study has assessed this parameter before and after a nasal desobstruction surgery.

The aim of the study is to evaluate the effect of nasal desobstruction surgery (septoplasty, septorhinoplasty or total ethmoidectomy) on sleep quality, assessed by the variation of the objective paraclinical criteria WASO, in patients presenting with sleep disorders and severe nasal obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic severe nasal obstruction of inflammatory (PNS) and/or morphological (symptomatic septal deviation) requiring surgical management
* NOSE > 9/20
* BMI < 30 kg/m2
* Over 18 years of age
* Pittsburgh Sleep Quality Index (PSQI) greater than or equal to 5

Exclusion Criteria:

* Patients with other sleep or wakefulness disorders: central sleep apnea syndromes, central hypersomnias including narcolepsy, parasomnia, restless legs syndrome and periodic leg movements.
* Craniofacial developmental abnormalities that may be responsible for OSA (retrognathia, endognathia, micro-mandibula, ogival palate, other occlusive disorder)
* Other identifiable obstructive site of the upper airways: tonsillar hypertrophy grade 3 and 4, macroglossia, unoperated vegetation hypertrophy, Mallampati score III or IV.
* Suspicion of anxiety or depressive disorder on the Hospital Anxiety and Depression scale (HAD) screening scale with H>10 and/or A>10.
* Use of psychotropic drugs or other respiratory depressant substances (morphine, chronic alcohol use, etc.)
* Night worker
* Other chronic rhinitis and rhinosinusitis
* Uncontrolled allergies
* Uncontrolled chronic respiratory disease
* Pregnancy
* Breastfeeding
* Subjects referred to in articles L.1121-5 to L.1121-8 and L.1122-1-2 of the public health code (e.g.: protected adults, people in emergency situations, people unable to give their personal consent etc...)
* Impossibility to understand the instructions and to answer in French
* impossibility to participate in the entire study
* no coverage by Social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
Wake after sleep onset | 6 months after inclusion (M0)
  Wake after sleep onset in minutes

SECONDARY OUTCOMES:
Total Sleep time | Change from baseline (M0) and 4 month after surgery (M6)
  Total sleep time in minutes
Time in bed | Change from baseline (M0) and 4 month after surgery (M6)
  Time in bed in minutes
Sleep latency | Change from baseline (M0) and 4 month after surgery (M6)
  Duration of time in minutes from turning the light off to falling asleep
Sleep efficiency | Change from baseline (M0) and 4 month after surgery (M6)
  ratio of total sleep time to time in bed
Pittsburgh Sleep Quality Index | Change from baseline (M0) and 4 month after surgery (M6)
  Index from 0 (meaning that there are no difficulties) to 21 (indicating major difficulties) about quality of sleep (the lowest is the index the better is the quality of sleep)
Pichot Qualitative Fatigue Scale score | Change from baseline (M0) and 4 month after surgery (M6)
  the Fatigue os measured by Pichot Qualitative Fatigue Scale witch is a 8-items self-administered questionnaire asking about fatigue.
  A 5-points scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 32.
  A score above 22 means an excessive state of fatigue
Epworth Sleepiness Scale (ESS) score | Change from baseline (M0) and 4 month after surgery (M6)
  Sleepiness complaints with ESS questionnaire. The ESS score can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life, or their 'daytime sleepiness'.
Insomnia Severity Index | Change from baseline (M0) and 4 month after surgery (M6)
  The Insomnia Severity Index is a 7-item self-administered questionnaire asking about difficulties sleeping and thoughts and worries about sleep.
  A 5-point scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28.
  The total score is interpreted as follows:
  absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Nasal obstruction scale | Change from baseline (M0) and 4 month after surgery (M6)
  Nasal Respiratory complaints measured by Nasal Obstruction Symptom Evaluation (NOSE questionnaire) The NOSE Scale is a 5-items self-administered questionnaire asking nose obstruction.
  A 5-points scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 20.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No